CLINICAL TRIAL: NCT02133014
Title: The Study of Laparoscopic-assisted Percutaneous Catheter-directed Drainage to Treat Early Severe Acute Pancreatitis in Chinese Population.
Brief Title: The Study of Laparoscopic-assisted Percutaneous Catheter-directed Drainage to Treat Early Severe Acute Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fanyingfang1
Record Dates: First submitted 2014-04-28; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Pancreatitis, Acute Necrotizing
Keywords: pancreatitis; laparoscopic; drainage; surgery
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatitis | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- surgical operation therapy (Experimental): Using the method of laparoscopic-assisted percutaneous catheter drainage of SAP.After the surgery,patient's cavity are continuously douched by catheter using 0.5% 5-fluorouracil normal saline.
  Interventions: Procedure: laparoscopic-assisted percutaneous catheter drainage; Drug: 0.5% 5-fluorouracil normal saline
- conventional therapy (No Intervention): using the method of conventional conservative therapy without surgical management.

INTERVENTIONS:
Procedure: laparoscopic-assisted percutaneous catheter drainage — Removing necrotic pancreatic organizations and putting the catheter around the region of pancreas.After the surgery,patient's cavity are continuously douched by catheter using 0.5% 5-fluorouracil normal saline
  Other Names: surgical therapy
  Arms: surgical operation therapy
Drug: 0.5% 5-fluorouracil normal saline — On the one hand,0.5% 5-fluorouracil normal saline directly inhibit DNA synthesis of pancreatic acinar cells which result in the synthesis of amylopsin of and trypsase is restrained.On the other hand,it can induce pancreatic cells apoptosis and alleviate pancreatic necrosis.
  Other Names: 5-FU; f5U
  Arms: surgical operation therapy

SUMMARY:
The purpose of this study is to analyze the effect of laparoscopic-assisted percutaneous catheter drainage of early SAP(severe acute pancreatitis).We are going to select 60 cases SAP patients from April 2014 to April 2015 who carry on the treatment in our hospital,and divide into the experimental group and control group under respect the wishes of patient in the case.The experimental group use the method of laparoscopic-assisted percutaneous drainage to carry on the treatment,the control group patients use conventional conservative therapy to carry on the treatment.Contrastive analyze two groups of patients clinical care effects.

Research hypothesis:according to compare the mortality,the incidence of complications ,hospital stay and other research indicators of two groups .It is supposed that the research indicators of experimental group are lower than the control group ,difference was statistically significant(P<0.05).We can draw the conclusion that the method of laparoscopic-assisted percutaneous catheter drainage of early SAP is useful and deserve to be promoted on clinical.

DETAILED DESCRIPTION:
According to the unified inclusion and exclusion criteria,We are going to select 60 cases SAP patients who carry on the treatment in our hospital from April 2014 to April 2015,and divide into the experimental group and control group under respect the wishes of patients.

The experimental group use the method of laparoscopic-assisted percutaneous catheter-directed drainage of SAP.According to different causes,.For patients with simple gallbladder stones,it is going to carry out by laparoscopic cholecystectomy or cholecystotomy.For patients with both gallbladder and common bile duct stones,common bile duct exploration is performed.Removing necrotic pancreatic organizations and putting the catheter around the region of pancreas.After the surgery,patient's cavity are continuously douched by catheter using 0.5% 5-fluorouracil normal saline.The postoperation therapeutic program is same as the control group.

The control group use the method of conventional conservative therapy without surgical management,the principles of treatment include:(1)fasting,insert gastric tube,gastrointestinal decompression;(2)complement of blood volume,keeping water ,electrolyte and acid base balance;(3)inhibiting pancreatic enzyme and acid secretion;(4)using broad-spectrum antibiotic at the early phase;(5)improving microcirculation,dextrans and FuFangdanshen by IV;(6)early parenteral nutrition;(7)treatment by chinese herbs;(8)strengthen the function of important organs.

Contrastive analyse two groups of patient's mortality,the incidence of complications,hospital stay,laboratory tests and other research indicators.

ELIGIBILITY:
Inclusion Criteria:Possessing the clinical performance and biochemical changes of acute pancreatitis,as well as one of the following items:

* organ dysfunction(one organ or multiple organs)
* local complications(pancreatic necrosis;pancreatic abscess;pancreatic pseudocyst);Ronson score of ≥3;
* APACHE-Ⅱscore of ≥8;
* Balthazar CT grade D or grade E.

Exclusion Criteria:

* mild acute pancreatitis;
* chronic acute pancreatitis;
* on admission has received surgical treatment;
* pregnant and lactating women ;combined with heart,lung,liver,kidney severe primary disease;psychopath;
* malignant tumor
* immunocompromised state.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
mortality | one year

SECONDARY OUTCOMES:
the incidence of local Complications | within the first 30 days (plus or minus 3 days) after surgery
  the local complications include:pancreatic necrosis,pancreatic abscess,pancreatic pseudocyst etc.

OTHER OUTCOMES:
hospital stay | participants will be followed for the duration of hospital stay, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fan y fang, Prof., Principal Investigator — Department of Hepatobiliary Surgery(I),Zhujiang Hospital
Locations (1):
- Department of Hepatobiliary Surgery(I),Zhujiang Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Echenique AM, Sleeman D, Yrizarry J, Scagnelli T, Guerra JJ Jr, Casillas VJ, Huson H, Russell E. Percutaneous catheter-directed debridement of infected pancreatic necrosis: results in 20 patients. J Vasc Interv Radiol. 1998 Jul-Aug;9(4):565-71. doi: 10.1016/s1051-0443(98)70323-9. PMID 9684824